CLINICAL TRIAL: NCT03829462
Title: A Randomized Phase III Trial Assessing a Regorafenib-irinotecan Combination (REGIRI) Versus Regorafenib Alone in Metastatic Colorectal Cancer Patients After Failure of Standard Therapies, According to the A/A Genotype of Cyclin D1
Brief Title: Assessing a Regorafenib-irinotecan Combination Versus Regorafenib Alone in Metastatic Colorectal Cancer Patients
Acronym: NEXT-REGIRI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2018-01 NEX
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: REGIRI; regorafenib; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan + regorafenib (REGIRI) (Experimental): irinotecan (180 mg/m2) at day1 of each cycle + regorafenib (160 mg/day) from day 2 to day 8
  Interventions: Drug: Regorafenib; Drug: Irinotecan
- regorafenib (Active Comparator): Regorafenib (160 mg/day) for 3 weeks followed by 1 week off
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — regorafenib tab 40 mg i.e 160 mg/day
Drug: Irinotecan — irinotecan 120 mg/m2 cycle 1, 150 mg/m2 cycle 2, 180 mg/m2 cycle 3 and more
  Arms: Irinotecan + regorafenib (REGIRI)

SUMMARY:
Patients with metastatic colorectal cancer (mCRC) who have received all approved standard treatments (except Regorafenib and Lonsurf) no longer have treatment options available while maintaining a good performance status which would allow them to receive a new treatment

DETAILED DESCRIPTION:
A Phase II randomized trial compared Nexiri (Nexavar® + Irinotecan) vs irinotecan or versus Sorafenib (Nexavar®). The patients treated with Irinotecan or Sorafenib alone could receive NEXIRI combination after progression (crossover to Nexiri).

Regorafenib, which is an oral signal deactivation agent with a chemical structure very similar to Sorafenib, is a standard treatment in heavily pretreated mCRC patients since the results of CORRECT study which compared Regorafenib to placebo on overall survival.

Sorafenib isn't approved in mCRC so the objective of this NEXT-REGIRI trial is compared REGIRI combination (Regorafenib-Irinotecan) to Regorafenib alone in a phase III trial in patients in progression after having received all standard treatments and bearing genotype A/A of cyclin D1. The study's hypothesis is that regorafenib could have effects similar to those of sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedures
* Male or female ≥ 18 years of age
* Histological documentation of adenocarcinoma of the colon or rectum
* Patients with metastatic colorectal cancer
* Progression during or within 3 months following the last administration of approved standard therapies, which must include a fluoropyrimidine (or raltitrexed), oxaliplatin, irinotecan, anti Vascular endothelial growth factor (VEGF) therapy and an anti Epithelial Growth Factor Receptor (EGFR) therapy (for RAS wild-type tumors)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Life expectancy of at least 3 months
* Patients with A/A cycline D1 (CCND1) genotype of rs603965 CCND1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: Amylase and lipase ≤1.5 x Upper Limit Normal (ULN),Total bilirubin ≤ 1.5 x ULN,Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer), Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5.0 x ULN for patients with liver involvement for their cancer and/or have bone metastases), Platelet count ≥ 100,000/mm3; Hemoglobin (Hb) ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥ 1,500/ mm3. Transfusion to meet the inclusion criterion, Serum creatinine ≤ 1.5 x ULN
* International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant, e.g., heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care
* Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment
* Women of childbearing potential and men must agree to use adequate contraception before entering the study until at least respectively 7 months and 4 months after the last study drug administration of Regorafenib and respectively 6 months and 3 months after the last study drug administration of Irinotecan. The investigator or a designated associate is requested to advise the patient on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.

Exclusion Criteria:

* Patients with A/G or G/G cycline d1 (CCND1) genotype of rs603965 CCND1
* Prior treatment with regorafenib or sorafenib
* Prior treatment with TAS 102
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of study drug
* Congestive heart failure ≥ New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Myocardial infarction less than 6 months before start of study drug
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension. (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE V5.0 Grade 2 dyspnea)
* Ongoing infection > Grade 2 NCI-CTCAE V5.0
* Known history of human immunodeficiency virus (HIV) infection
* Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Patients with seizure disorder requiring medication
* History of organ allograft
* Patients with evidence or history of any bleeding diathesis, irrespective of severity
* Any hemorrhage or bleeding event ≥ NCI-CTC V5.0 Grade 3 within 4 weeks prior to the start of study medication
* Non-healing wound, ulcer, or bone fracture
* Dehydration NCI-CTCAE V5.0 Grade ≥ 1
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Any illness or medical conditions that are unstable or could
* jeopardize the safety of the subject and his/her compliance in the study
* Persistent proteinuria of NCI-CTCAE V5.0 Grade 3 (> 3.5g/24 hours)
* Patients unable to swallow oral medications
* Any malabsorption condition
* Chronic inflammatory bowel disease and / or bowel obstruction
* Unresolved toxicity higher than NCI-CTCAE V.5.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neurotoxicity ≤ Grade 2
* Concomitant participation or participation within the last 30 days in another clinical trial
* Systemic anticancer therapy during this trial or within 4 weeks before randomization
* Concomitant intake of st John's wort
* Live attenuated vaccines are prohibited 10 days before the treatment, during the treatment and 6 months after the termination of treatment
* History of gastrointestinal fistula or perforation
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to study inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (11):
- France (11):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - Centre François Baclesse, Caen, Basse-Normandie
  - Hôpital Pontchaillou, Rennes, Ile Et Vilaine
  - Hôpital Robert Debré, Reims, Marne
  - Institut Godinot, Reims, Marne
  - Hôpital Saint-Jean, Perpignan, Pyrénées-orientales
  - Centre Léon Bérard, Lyon, Rhône
  - Hôpital privé Jean Mermoz, Lyon, Rhône
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - CRLC Val d'Aurelle-Paul Lamarque, Montpellier
  - Hôpital Européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan, the clinical study report and the analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Access to study data upon written detailed request sent to Institute of Montpellier Cancer after publication.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Samalin E, Bouche O, Thezenas S, Francois E, Adenis A, Bennouna J, Taieb J, Desseigne F, Seitz JF, Conroy T, Galais MP, Assenat E, Crapez E, Poujol S, Bibeau F, Boissiere F, Laurent-Puig P, Ychou M, Mazard T. Sorafenib and irinotecan (NEXIRI) as second- or later-line treatment for patients with metastatic colorectal cancer and KRAS-mutated tumours: a multicentre Phase I/II trial. Br J Cancer. 2014 Mar 4;110(5):1148-54. doi: 10.1038/bjc.2013.813. Epub 2014 Jan 9. PMID 24407191
- [Background] Lu F, Gladden AB, Diehl JA. An alternatively spliced cyclin D1 isoform, cyclin D1b, is a nuclear oncogene. Cancer Res. 2003 Nov 1;63(21):7056-61. PMID 14612495
- [Background] Alt JR, Cleveland JL, Hannink M, Diehl JA. Phosphorylation-dependent regulation of cyclin D1 nuclear export and cyclin D1-dependent cellular transformation. Genes Dev. 2000 Dec 15;14(24):3102-14. doi: 10.1101/gad.854900. PMID 11124803
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 11 academic medical centers between March 2019 (first patient screened but non randomized) and august 2024.The first patient was randomized on September 18, 2019 and the last patient was randomized in march 2024.
Pre-assignment Details: After enrollment, a screening was carried out according to the polymorphism (A870A rs603965) of cyclin D1, a protein involved in cell cycle regulation.Of 377 enrolled patients, 66 patients met selection criteria and were randomized to the study.In the protocol, we had planned to randomize 78 patients, but we had also specified that endpoints could be analyzed as soon as 55 events (deaths) were reached (i.e when one of the two is reached first).
Period: Overall Study
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Started | 33 | 33
Per Protocol Population at 8 Weeks With a Evaluation by CT Scan | 27 | 29
Completed | 27 | 29
Not Completed | 6 | 4
Not completed — No tumoral evaluation due to progression disease | 6 | 3
Not completed — No treatment due to progression disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 38
  >=65 years | 16 | 12 | 28
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 78] | 64 [37 to 75] | 64 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 21 | 15 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 33 | 66
Region of Enrollment [Number; unit: participants]
  France | 33 | 33 | 66
RAt Sarcoma virus (RAS) Status [Number; unit: participants] — Ras is a family of proteins with a protooncogenic role. Approximately, one in two human colorectal tumors has a mutation in this gene.
  Patients with a mutant RAS gene cannot receive Cetuximab treatment and cetuximab-like treatment due to treatment resistance.
  participants
    wild RAS | 15 | 14 | 29
    Mutant RAS | 18 | 19 | 37
Genotype of cycline D1 (polymorphism A/A) [Number; unit: participants] — Cyclin D1 is a protein involved in cell cycle regulation and transcription. Our hypothesis is that patients with the Cycline D1 polymorphism A/A could have a better response with the REGIRI (Regorafenib + Irinotecan) combination on overall survival compared with the two other genotypes A/G and G/G.
  participants | 33 | 33 | 66
Microsatellite Stability (MSS) Status [Number; unit: participants] — The patients with a phenotype of microsatellite instability has a DNA mismatch repair system deficiency.
  participants
    Missing | 4 | 4 | 8
    Mutant MSS (microsatellite stability biomarker) | 29 | 29 | 58
v-RAF murine sarcoma viral oncogene homolog B (BRAF) Status [Number; unit: participants] — This gene encodes a protein belonging to the RAF family of serine/threonine protein kinases. Protooncogenic protein that helps transmit chemical signals from outside the cell to the cell nucleus. This protein regulates cell growth and division.
  participants
    Wild BRAF | 29 | 23 | 52
    Mutant BRAF | 1 | 1 | 2
    Missing | 3 | 9 | 12
World Health Organization (WHO) status performance index [Number; unit: participants] — The World Health Organization (WHO) performance status is a scale used to assess the general well-being and activities of daily life of a cancer patient.
  Scale 0 to 5 (0= the best general well-being, 5=death).
  participants
    WHO=0 | 10 | 18 | 25
    WHO=1 | 23 | 18 | 41
MALE WEIGHT [Median (Full Range); unit: KG] — Population: Of 33 patients randomized to arm A, 21 are men. Of 33 patients randomized to arm B, 15 are men.
  KG
    number analyzed (Participants) | 21 | 15 | 36
    (all) | 75.2 [50 to 94] | 82.6 [51 to 107] | 77.5 [50 to 107]
FEMALE WEIGHT [Median (Full Range); unit: KG] — Population: Of 33 patients randomized to arm A, 12 are women. Of 33 patients randomized to arm B, 18 are women.
  KG
    number analyzed (Participants) | 12 | 18 | 30
    (all) | 56.1 [43.2 to 93] | 65.2 [39 to 99] | 61.3 [39 to 99]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m²] | 24.4 [17.9 to 33.3] | 25.3 [17.3 to 37.5] | 24.6 [17.3 to 37.5]
Significant medical and surgical history [Number; unit: participants]
  no | 3 | 6 | 9
  yes | 30 | 27 | 57
Ongoing signs and symptoms [Number; unit: participants]
  no | 11 | 10 | 21
  yes | 22 | 23 | 45
Location of primary tumor [Number; unit: participants]
  Right colon | 8 | 7 | 15
  Left colon | 9 | 7 | 16
  transverse colon | 1 | 3 | 4
  Recto-sigmoid junction | 6 | 7 | 13
  Rectum | 9 | 9 | 18
Tumor (T) from TNM classification given by pathologist [Number; unit: participants] — The TNM classification is determined by pathologist when he analyzes the colonic or rectal tumor.
  T for tumor : Tis (in situ carcinoma) better outcome and T4 (tumor perforating the peritoneum) worse outcome.
  N for number of nodes invaded : (N0 indicates the absence of lymph node invasion by tumor cells, better outcome, N1 (1 to 3 lymph nodes invaded) and N2 (more 4 lymph nodes invaded, worse outcome).
  M for presence of metastasis : M0 absence of metastasis, better outcome ; M1 presence, worse outcome.
  participants
    T1 (tumor invading the submucosa) | 1 | 0 | 1
    T2 (tumor invading the muscularis) | 0 | 3 | 3
    T3 (tumor invading the subserosa) | 17 | 7 | 24
    T4 (tumor perforating the peritoneum or invading other organs) | 7 | 13 | 20
    Tis (in situ carcinoma) | 0 | 1 | 1
    Tx (unknown) | 8 | 9 | 17
pN (node) from TNM classification given by pathologist [Number; unit: participants] — The TNM classification is determined by pathologist when he analyzes the colonic or rectal tumor.
  T for tumor : Tis (in situ carcinoma) better outcome and T4 (tumor perforating the peritoneum) worse outcome.
  N for number of nodes invaded : (N0 indicates absence of lymph node invasion by tumor cells, better outcome, N1 (1 to 3 lymph nodes invaded) and N2 (> 4 lymph nodes invaded, worse outcome).
  M for presence of metastasis : M0 absence, better outcome ; M1 presence, worse outcome.
  participants
    pN0 (no lymph node invaded) | 3 | 7 | 10
    pN1 (1 to 3 lymph nodes invaded) | 12 | 7 | 19
    pN2 (> 4 lymph nodes invaded) | 8 | 9 | 17
    pNx (unknown) | 10 | 10 | 20
pM from TNM classification given by pathologist [Number; unit: participants] — The TNM classification is determined by pathologist when he analyzes the colonic or rectal tumor.
  T for tumor : Tis (in situ carcinoma) better outcome and T4 (tumor perforating the peritoneum) worse outcome.
  N for number of nodes invaded : (N0 indicates absence of lymph node invasion by tumor cells, better outcome, N1 (1 to 3 lymph nodes invaded) and N2 (> 4 lymph nodes invaded, worse outcome).
  M for presence of metastasis : M0 absence, better outcome ; M1 presence, worse outcome.
  participants
    M0 (absence of metastasis) | 6 | 4 | 10
    M1 (presence of metastasis) | 22 | 20 | 42
    MX (unknown) | 5 | 9 | 14
lymph-node removal [Number; unit: participants] — Bad prognosis if nodes are not removed.
  participants
    no | 14 | 17 | 31
    yes | 19 | 16 | 35
Number of patients with nodes removed [Count of Participants; unit: Participants] — ARM A :
  19 patients with lymph nodes removal 14 patients without lymph nodes removal
  ARM B :
  16 patients with lymph nodes removal 17 patients without lymph nodes removal
  Participants | 19 | 16 | 35
Number of patients with invaded nodes [Count of Participants; unit: Participants] — ARM A :
  19 patients with lymph nodes invaded and 14 patients without lymph nodes invaded
  ARM B :
  16 patients with lymph nodes invaded and 17 patients without lymph nodes invaded
  Participants | 19 | 16 | 35
Type of adenocarcinoma [Number; unit: participants] — The type of adenocarcinoma is determined by the pathologist when he analyzes the colonic or rectal tumor.
  participants
    Colloide adenocarcinoma | 2 | 3 | 2
    LIEBERKUHNIEN adenocarcinoma | 27 | 33 | 60
    Other adenocarcinoma | 4 | 0 | 4
Number of metastatic sites [Number; unit: participants]
  1 metastatic site | 18 | 18 | 36
  2 metastatic sites | 11 | 13 | 24
  3 metastatic sites | 3 | 2 | 5
  4 metastatic sites | 1 | 0 | 1
Location of metastases [Number; unit: participants]
  Lung | 12 | 14 | 26
  Liver | 25 | 27 | 52
  Peritoneum | 10 | 3 | 13
  Distant lymph nodes | 4 | 4 | 8
  Other (ovaries, adrenal glands, peritoneum) | 2 | 2 | 4
Previous surgery number [Number; unit: participants]
  0 | 8 | 8 | 16
  1 | 13 | 9 | 22
  2 | 12 | 12 | 24
  3 | 0 | 3 | 3
  4 | 0 | 1 | 1
Carcinoembryonic antigen (CEA) Biomarker [Median (Full Range); unit: ng/ml] — Blood CEA levels are often higher in the presence of colorectal cancer. CEA quantitative analysis has important prognostic value in colon cancer and in the Post-treatment monitoring of colorectal cancer.
  ng/ml | 57.1 [3.1 to 1108] | 46.1 [3.5 to 7916.6] | 52.75 [3.1 to 7916.6]
Carbohydrate Antigen 19-9 (CA 19-9) Biomarker [Median (Full Range); unit: U/ml] — CA-19-9 levels are often higher in the presence of colorectal cancer. CA19-9 quantitative analysis has important prognostic value in colon cancer and in the Post-treatment monitoring of colorectal cancer.
  U/ml | 98 [0 to 297000] | 68 [1 to 9922.5] | 89 [0 to 297000]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: Up to 36 months
Population: Population per-protocol
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 27 | 29
Month | 9 [6.1 to 14.5] | 5.5 [3.8 to 13.4]
Statistical Analysis 1: Comparison: Irinotecan + Regorafenib (REGIRI) vs Regorafenib; To show an increase of median overall survival from 7 to 15 months (30% to 57% rates, respectively), with a HR=0.47 and a power of 80% and alpha=5%, 55 events are required for the 78 patients to be randomized considering 15% additional patients for lost to follow-up; Test type: Superiority; p = 0.5334, Log Rank — The threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.7 to 1.98]
Statistical Analysis 2: Comparison: Irinotecan + Regorafenib (REGIRI); Test type: Superiority; p = 0.8894, Chi-squared; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.59 to 1.82]

2. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 36 months
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 33 | 33
month | 3.6 [2 to 4.2] | 1.9 [1.8 to 2.1]
Statistical Analysis 1: Comparison: Irinotecan + Regorafenib (REGIRI) vs Regorafenib; Test type: Superiority; p = 0.1104, Log Rank; The threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.4 to 1.11]
Statistical Analysis 2: Comparison: Irinotecan + Regorafenib (REGIRI); Test type: Superiority; p = 0.1165, Chi-squared; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.4 to 1.11]

3. Secondary Outcome: Time to Deterioration
Time Frame: Up to 36 months
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 33 | 33
month | 4.6 [3.6 to 5] | 2.1 [1.4 to 3]
Statistical Analysis 1: Comparison: Irinotecan + Regorafenib (REGIRI) vs Regorafenib; Test type: Superiority; p = 0.2425, Log Rank — The threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.26 to 1.42]
Statistical Analysis 2: Comparison: Irinotecan + Regorafenib (REGIRI); Test type: Superiority; p = 0.2519, Chi-squared; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.26 to 1.42]

4. Secondary Outcome: Number of Participants With Disease Control Rate
Time Frame: Through study completion, up to 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 27 | 29
Participants | 20 | 8
Statistical Analysis 1: Comparison: Irinotecan + Regorafenib (REGIRI); Test type: Superiority; p = 0.001, Fisher Exact; Percent difference = 46.5

5. Secondary Outcome: Number of Patients With an Objective Response Rate
Time Frame: Through treatment completion, up to 14 months
Population: Population Per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 27 | 29
Participants | 2 | 0
Statistical Analysis 1: Comparison: Irinotecan + Regorafenib (REGIRI); Test type: Superiority; p = 0.001, Fisher Exact; Percent difference = 7.4

6. Secondary Outcome: Assessment of Adverse Events by Using the NCI-CTCAE Version 5.0 Scale (Grade Max Per Patient)
Time Frame: Up to 36 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 33 | 32
Participants
  Grade 1 | 4 | 2
  Grade 2 | 13 | 8
  Grade 3 | 9 | 21
  Grade 4 | 4 | 1
  Grade 5 | 3 | 0

7. Secondary Outcome: Quality of Life Questionnaire
Description: The Quality of Life questionnaire (QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients.
  The QLQ-C30 incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia and diarrhea) and perceived financial impact of the disease. Score 0 to 100 for all subscales.
  * Functional scale : 0 the worst outcome, 100 is the best outcome,
  * Symptomatic scale : 0 the best outcome, 100 is the worst outcome Global functioning measures how much a person's symptoms affect their day-to-day life and role functioning assesses a patient's ability to perform daily activities, leisure time activities, and work on a scale of 0 to 100 (0 the worst outcome and 100 the best outcome).
Time Frame: Questionnaire is assessed until 16 weeks (baseline, 8 weeks and 16 weeks)
Population: The number of patients differs from the ITT population because some patients have not completed the questionnaires. Therefore the analysis is carried out on a smaller population, those who responded to the questionnaires. The table below shows the median scores of scales ranging from 0 to 100.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
Number analyzed (Participants) | 21 | 16
Units on a scale
  GLOBAL HEALTH STATUS AT BASELINE | 63 [25 to 83.33] | 67 [16.67 to 100]
  PHYSICAL FUNCTIONING AT BASELINE | 93 [46.67 to 100] | 75 [16.67 to 100]
  ROLE FUNCTIONING AT BASELINE | 100 [0 to 100] | 75 [16.67 to 100]
  EMOTIONAL FUNCTIONING AT BASELINE | 83 [25 to 100] | 92 [25 to 100]
  COGNITIVE FUNCTIONING AT BASELINE | 83 [33.33 to 100] | 100 [50 to 100]
  SOCIAL FUNCTIONING AT BASELINE | 100 [33.33 to 100] | 75 [33.33 to 100]
  ASTHENIA AT BASELINE | 33 [0 to 77.78] | 33 [0 to 88.89]
  NAUSEA AND VOMITING AT BASELINE | 0 [0 to 66.67] | 0 [0 to 100]
  PAIN AT BASELINE | 33 [0 to 100] | 17 [0 to 100]
  DYSPNEA AT BASELINE | 0 [0 to 66.67] | 17 [0 to 66.67]
  INSOMNIA AT BASELINE | 33 [0 to 100] | 33 [0 to 100]
  APPETITE LOSS AT BASELINE | 0 [0 to 100] | 17 [0 to 100]
  DIARRHEA AT BASELINE | 0 [0 to 100] | 17 [0 to 66.67]
  FINANCIAL DIFFICULTIES AT BASELINE | 0 [0 to 66.67] | 0 [0 to 33.33]
  GLOBAL HEALTH STATUS AT 8 WEEKS | 67 [33.33 to 83.33] | 50 [33.33 to 83.33]
  PHYSICAL FUNCTIONING AT 8 WEEKS | 87 [33.33 to 100] | 40 [33.33 to 80]
  ROLE FUNCTIONING AT 8 WEEKS | 83 [33.33 to 100] | 33 [0 to 66.67]
  EMOTIONAL FUNCTIONING AT 8 WEEKS | 83 [41.67 to 100] | 83 [33.33 to 100]
  COGNITIVE FUNCTIONING AT 8 WEEKS | 83 [50 to 100] | 100 [16.67 to 100]
  SOCIAL FUNCTIONING AT 8 WEEKS | 83 [0 to 100] | 83 [16.67 to 100]
  ASTHENIA AT 8 WEEKS | 33 [0 to 100] | 78 [22.22 to 100]
  NAUSEA AND VOMITING AT 8 WEEKS | 0 [0 to 33.33] | 0 [0 to 83.33]
  PAIN AT 8 WEEKS | 33 [0 to 100] | 67 [0 to 100]
  DYSPNEA AT 8 WEEKS | 33 [0 to 100] | 33 [0 to 100]
  INSOMNIA AT 8 WEEKS | 0 [0 to 100] | 33 [0 to 100]
  APPETITE LOSS AT 8 WEEKS | 0 [0 to 100] | 33 [0 to 100]
  DIARRHEA AT 8 WEEKS | 33 [0 to 100] | 33 [0 to 100]
  FINANCIAL DIFFICULTIES AT 8 WEEKS | 0 [0 to 66.67] | 0 [0 to 33.33]
  GLOBAL HEALTH STATUS AT 16 WEEKS | 58 [16.67 to 100] | 58 [41.67 to 66.67]
  PHYSICAL FUNCTIONING AT 16 WEEKS | 80 [53.33 to 100] | 63 [53.33 to 80]
  ROLE FUNCTIONING AT 16 WEEKS | 67 [33.33 to 100] | 67 [50 to 83.33]
  EMOTIONAL FUNCTIONING AT 16 WEEKS | 75 [41.67 to 100] | 79 [75 to 83.33]
  COGNITIVE FUNCTIONING AT 16 WEEKS | 100 [66.67 to 100] | 92 [83.33 to 100]
  SOCIAL FUNCTIONING AT 16 WEEKS | 67 [33.33 to 100] | 75 [66.67 to 100]
  ASTHENIA AT 16 WEEKS | 44 [0 to 88.89] | 44 [22.22 to 66.67]
  NAUSEA AND VOMITING AT 16 WEEKS | 0 [0 to 100] | 0 [0 to 100]
  PAIN AT 16 WEEKS | 33 [0 to 66.67] | 8 [0 to 66.67]
  DYSPNEA AT 16 WEEKS | 0 [0 to 66.67] | 33 [0 to 33.33]
  INSOMNIA AT 16 WEEKS | 33 [0 to 66.67] | 50 [0 to 100]
  APPETITE LOSS AT 16 WEEKS | 0 [0 to 100] | 33 [0 to 66.67]
  DIARRHEA AT 16 WEEKS | 33 [0 to 100] | 33 [0 to 66.67]
  FINANCIAL DIFFICULTIES AT 16 WEEKS | 0 [0 to 66.67] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the baseline up to one month after the last cycle of chemotherapy, up to 36 months. All-Cause Mortality was assessed through study completion, up to 36 months.
Arm/Group | Irinotecan + Regorafenib (REGIRI) | Regorafenib
All-Cause Mortality (participants affected / at risk) | 32/33 | 27/33
Serious Adverse Events (participants affected / at risk) | 21/33 | 20/33
Other Adverse Events (participants affected / at risk) | 33/33 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan + Regorafenib (REGIRI) (N=33) | Regorafenib (N=33)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coloanal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Occlusive syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stenosis of coloretal anastomosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Deterioration in general condition (General disorders) | 3 (3) | 4 (4)
Fever (General disorders) | 2 (2) | 1 (1)
Stroke (Cardiac disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3)
Catheter infection (Infections and infestations) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Arterial hypertension (Vascular disorders) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis due to digestive perforation (Infections and infestations) | 1 (1) | 0 (0)
Left superior member hemiparesis (General disorders) | 1 (1) | 0 (0)
Malposition of Hubert needle (Surgical and medical procedures) | 1 (1) | 0 (0)
Maculopapular exanthema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 2 (2) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan + Regorafenib (REGIRI) (N=33) | Regorafenib (N=33)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (21) | 1 (2)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Acneiform rash (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4)
Skin dryness (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 10 (15) | 13 (19)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (2)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 4 (5)
Dysgueusia (Nervous system disorders) | 2 (3) | 1 (1)
Insomnia (Nervous system disorders) | 1 (2) | 1 (2)
Peripheral neuropathy (Nervous system disorders) | 6 (10) | 6 (9)
Peripheral neuropathyneuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (4) | 1 (1)
Canker sore (Gastrointestinal disorders) | 0 (0) | 3 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (30) | 20 (50)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (1)
haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mucositis (Gastrointestinal disorders) | 3 (6) | 5 (6)
Nausea (Gastrointestinal disorders) | 15 (23) | 1 (1)
odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
rectorrhagia (Gastrointestinal disorders) | 2 (3) | 3 (4)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 6 (7)
Leucopenia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Neutropenia (Gastrointestinal disorders) | 6 (8) | 0 (0)
Thrombopenia (Blood and lymphatic system disorders) | 2 (3) | 7 (10)
Cholestasis (Gastrointestinal disorders) | 7 (8) | 2 (2)
Hepatic pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Right hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bones pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Sciatica pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Caruncle inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Running nose (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nose bleeding (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 9 (13)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Heat/cold sensation (Vascular disorders) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 3 (4) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Facial folliculatis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Urinary infection (Infections and infestations) | 0 (0) | 1 (1)
Right eye stye (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal skin superinfection (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 4 (5)
Alanine aminotransferase increased (Investigations) | 7 (10) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (7) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 12 (17) | 5 (7)
Lipase increased (Investigations) | 1 (2) | 4 (6)
Weight loss (Investigations) | 6 (7) | 6 (8)
Anastomosis stenosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Albumenia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 9 (12) | 10 (16)
Hyperkaliema (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cytolysis (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokaliema (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Deterioration general condition (General disorders) | 1 (1) | 5 (5)
Pain (General disorders) | 7 (9) | 16 (25)
Asthenia (General disorders) | 25 (37) | 19 (31)
Fever (General disorders) | 7 (10) | 7 (8)
Edema of the limbs (General disorders) | 2 (2) | 1 (1)
Inflammatory syndrome (General disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Voice alteration (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Epigastralgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Left ear deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Occlusion (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* In the protocol, we had planned to randomize 78 patients, but we had also specified that endpoints could be analyzed as soon as 55 events (deaths) were reached (i.e when one of the two is reached first). When inclusion ended, we continued to record deaths and obtained 59 events for 66 randomized patients i.e 33 patients randomized in each arm.
* There is no data on race or ethnicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT03829462/Prot_SAP_000.pdf